CLINICAL TRIAL: NCT06909201
Title: Hyperpolarized Xenon-129 Magnetic Resonance Imaging in Lung Cancer Patients Receiving Radiation Therapy for Investigating Radiation-response and Toxicity
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1200
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: High-Risk RP Patients (Experimental)
  Interventions: Drug: HP 129Xe MRI
- Arm B: Low-Risk RP Patients (Experimental)
  Interventions: Drug: HP 129Xe MRI
- Arm C: Healthy Volunteers (Negative Control) (Experimental)
  Interventions: Drug: HP 129Xe MRI

INTERVENTIONS:
Drug: HP 129Xe MRI — Gas delivery will be from a Tedlar bag

SUMMARY:
The goal of this clinical research study is to learn if novel type of imaging scan called HP 129Xe MRI can help doctors identify and predict common side effects of radiation therapy. Rather than contrast-enhanced MRIs, the tracer (129Xe) will be inhaled rather than injected.

The 129Xe tracer has not been FDA approved. Its use in this study is investigational.

DETAILED DESCRIPTION:
Primary Objectives:

To assess the association between imaging features on longitudinal HP 129Xe MRI and the development and severity of radiation pneumonitis resulting from radiation therapy for non-small cell lung cancer.

To determine if HP 129Xe MRI features, in conjunction with a given patient's radiation treatment plan, can predict radiation pneumonitis development and severity.

Secondary Objectives:

Optimize HP 129Xe MRI acquisition techniques.

To determine if HP 129Xe MRI can pre-emptively detect radiation pneumonitis prior to symptom presentation.

Compare changes in HP 129Xe MRI metrics to CT-based ventilation metrics over the course of radiation therapy.

To identify pulmonary regions more susceptible to radiation damage.

To develop alternative radiation treatment plans, based on HP 129Xe MRI features of lung function, that may prevent radiation pneumonitis development and compare to standard-of-care treatment plans.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control cohort:

   1. Able to consistently hold breath for 10-12 seconds
   2. No history of any pulmonary disorders (i.e., asthma, COPD, lung cancer, etc.)
   3. Able to undergo MRI examination
   4. At least 18 years of age
2. Lung cancer patient cohort:

   1. Biopsy proven diagnosis of lung cancer
   2. Receiving photon- or proton-based external beam radiotherapy as a part of treatment
   3. Able to undergo MRI examination
   4. Will receive follow-up at University of Texas MD Anderson Cancer Center (UTMDACC)
   5. Able to consistently hold breath for 10-12 seconds
   6. Women and men with child-bearing potential agree to use adequate contraception prior to study entry and during the duration of study participation.
   7. Able to understand and willing to sign a written informed consent document
   8. At least 18 years of age

The effects of HP 129Xe MRI on the developing human fetus are unknown. For this reason and because radiotherapy is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Additionally, if female partners of male study participants become pregnant during study participation, the treating physician should be informed immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients unable to follow up at MD Anderson for routine clinical care
2. Inability or unwillingness to give informed consent
3. Relapsed disease or life expectancy less than 6 months at time of enrollment
4. Severe claustrophobia precluding MRI imaging active pulmonary infection
5. Pregnant women
6. Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Niedzielski, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org